CLINICAL TRIAL: NCT01289613
Title: Clinically Relevant Asymmetry of Bispectral Index During Anesthesia for ENT Surgery in Adults and Children
Brief Title: Clinically Relevant Asymmetry of Bispectral Index
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Axel Fudickar, Dr. med., University Hospital Schleswig-Holstein
Other Study IDs: USchleswig-Holstein
Record Dates: First submitted 2011-02-02; First posted 2011-02-04 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Reaction; Anesthesia
Keywords: Bispectral Index; Anesthesia; Asymmetry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children: Children
- Adults: Adults

SUMMARY:
BIS for monitoring depth of anesthesia is usually obtained unilaterally. Obtaining BIS bilaterally revealed side differences in previous studies. This study investigates the incidence of clinically relevant side differences of BIS during maintenance and emergence from anesthesia for ENT surgery in both adults and children.

DETAILED DESCRIPTION:
BIS was measured bilaterally in 42 adults and 46 children during ENT surgery under general anesthesia using two BIS-Monitors. Side differences of more than 10% were defined as BIS asymmetries. An increase of BIS of more than 10% from the value at the time of finishing anesthesia administration on only one side followed by movement after stimulation was defined as clinically relevant.

ELIGIBILITY:
Inclusion Criteria:Children and adults during anesthesia for ENT surgery -

Exclusion Criteria:Neurologic or psychiatric disease

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults during anesthesia for ENT surgery
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Movement reaction to external stimulation during emergence from anesthesia | 30 minutes
  After surgery, administration of propofol and remifentanil was stopped and the measurement of BIS was continued. BIS was noted every minute and on each occasion BIS exceeded 10% of the value at stopping the application of anesthetics on one or both sides. If such a 10% increase was observed, arousal and movement after external stimulation was examined by suction of the mouth.
  BIS asymmetry on only one side followed by movement reaction to external stimulation within a 60 seconds period was defined as clinically relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Fudickar, Dr., Principal Investigator — University Clinic Schleswig-Holstein, Campus Kiel
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Germany